CLINICAL TRIAL: NCT03901235
Title: Treatment of Refractory Crohn's Disease Lesions by Local Injection of Mesenchymal Stem Cells
Brief Title: MSC Intratissular Injection in Crohn Disease Patients
Acronym: MSC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Collaborators: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Edouard Louis, Prof, University of Liege
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJT1707P1
Record Dates: First submitted 2019-03-04; First posted 2019-04-03 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Efficacy and Safety

STUDY DESIGN:
Intervention Model Description: Non-controlled, non-randomized, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mesenchymal Stromal Cells (Experimental)
  Interventions: Biological: Mesenchymal Stromal Cells

INTERVENTIONS:
Biological: Mesenchymal Stromal Cells — Suspension of mesenchymal stromal cells for intratissular injection

SUMMARY:
The main objective is to assess the efficacy of local injection of MSC on the healing of refractory intestinal and perianal lesions in crohn disease. The second co-primary endpoint is safety.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age
* Signing the informed consent
* Diagnosis of Crohn Disease for more than 6 months
* Presence of at least one Crohn Disease lesion refractory to conventional therapies (azathioprine, 6-mercaptopurine or methotrexate) and to biologic treatments (anti-Tumor Necrosis Factor therapies, vedolizumab, or ustekinumab).
* Refractory lesion defined by (1) a stricture with a length of 2 to 5cm of the colon or the ileum accessible by ileocolonoscopy (i.e. a lesion identified during a colonoscopy with a lumen narrowing non passable by the colonoscope), (2) unhealed deep ulcer of the colon or the ileum accessible to ileocolonoscopy, or (3) actively draining perianal fistula(s).
* Twenty patients with stricture(s), 20 patients with unhealed deep ulcer(s), and 20 patients with an actively draining perianal fistula(s) will be included

Exclusion Criteria:

* Indication for immediate luminal surgery
* Intestinal obstruction
* Intra-abdominal fistulas or abscess
* Intestinal/colonic stricture or deep unhealed ulcer not accessible to ileocolonoscopy
* Undrained peri-anal abscess
* Pregnant women or planning pregnancy within one year
* Positive stool culture/toxin for clostridium difficile pathogen or other pathogens
* Renal failure (anuria, serious fluid overload, Glomerular Filtration Rate < 30 ml/min, dialysis) or hepatic failure (Fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin >3 mg/dL)
* documented human immunodeficiency virus infection; active hepatitis B, C, or tuberculosis
* an opportunistic infection within 6 months before screening or a serious infection in the previous 3 months
* malignancy within the past 5 years; or a history of lymphoproliferative disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with deep ulcer healing | Week 12
  Complete deep ulcer healing is defined by the disappearance of the ulcer; partial healing is defined by a decrease in the depth or the diameter of the ulcer.
Proportion of patients with stricture healing | Week 12
  Complete stricture healing is defined by the ability to pass the ileocolonoscope through the stricture; partial healing is defined by the increase in the diameter of the stricture.
Proportion of patients with complex perianal fistula healing | Week 12
  Complete complex perianal fistula healing is defined by the complete closure of the external fistula opening, no drainage upon gentle pressure, no abscess. And by looking at the size of the fistulous track, presence of collection, and gadolinium enhancement by MRI
Safety assessed by the incidence of treatment-emergent adverse events during the study period | from week 0 to week 48
  Assessment of the incidence of adverse and serious adverse events over the 48 weeks study period. Toxicity grade of adverse events is determined using the Common Terminology Criteria for Adverse Events (version 4.0). Relationship to the therapeutic procedure will systematically be assessed.

SECONDARY OUTCOMES:
Evolution of clinical disease activity index | week 0, 12 and 48
  Assess disease activity in Crohn's disease over 7 days using the Crohn's disease activity index
Evolution of Short health scale (quality of life) | week 0, 12 and 48
  min : 0 - max : 10 (worse)
Evolution of the Lemann Index (measuring cumulated intestinal damage in Crohn's disease) | week 0, 12 and 48
  which incorporates clinical, surgical, endoscopic, and imaging findings from all segments of the digestive tract into one composite score
Evolution of the " Group of Therapeutic Study of Inflammatory Disorders of the Digestive Tube" obstructive score for Crohn Disease strictures | weeks 0, 12 and 48
  Grade : from 0 to higher value 6

CONTACTS AND LOCATIONS:
Overall Officials: Edouard Louis, Prof, Principal Investigator — Centre Hospitalier Universitaire de Liege
Locations (1):
- CHU de Liège, Liège, Liège, Belgium